CLINICAL TRIAL: NCT04441879
Title: bBeAMom Trial: A Randomized Controlled Trial to Test the Effectiveness of a Cognitive-Behavioral Blended Intervention for Postpartum Depression in Portuguese Women
Brief Title: bBeAMom: Effectiveness of a Cognitive-Behavioral Blended Intervention for Postpartum Depression
Acronym: bBeAMom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Ana Fonseca, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bBeAMom/145563/2019; SFRH/BD/145563/2019 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Postpartum Depression
Keywords: Postpartum Depression; Cognitive-Behavioral Therapy; Web-Based Psychological Intervention; Blended intervention
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended intervention (Experimental): Women will receive a blended intervention (integrating face-to-face and online sessions) for the treatment of postpartum depression.
  Interventions: Behavioral: Be a Mom Coping with Depression
- Control (online intervention) (Active Comparator): Women will receive an online intervention (Be a Mom program).
  Interventions: Behavioral: Be a Mom

INTERVENTIONS:
Behavioral: Be a Mom Coping with Depression — Be a Mom Coping with Depression is a blended cognitive-behavioral intervention for the treatment of postpartum depression. It consists of 13 weeks of face-to-face and online sessions, each session targeting a specific thematic content, and providing participants with both information and specific therapeutic strategies (with a strong focus on cognitive-behavioral techniques) to address each thematic content.
  Arms: Blended intervention
Behavioral: Be a Mom — Be a Mom is an online intervention consisting of 6 modules, each one targeting a specific thematic content, and providing women with both information and specific therapeutic strategies (with a strong focus on cognitive-behavioral techniques) to address each thematic content. Women will receive biweekly phone calls from a psychologist between completion of each module to provide support.
  Arms: Control (online intervention)

SUMMARY:
Be a mom program (a web-based cognitive-behavioral intervention) is being tested in another clinical trial as a preventive intervention for postpartum depression (NCT03024645). However, given its effectiveness in reducing depressive symptoms among women presenting early-onset postpartum depressive symptoms, Be a Mom can also have potential as a postpartum depression complement treatment tool. The main goal of this research is to apply and evaluate the acceptability and effectiveness of a blended cognitive-behavioral intervention for the treatment of postpartum depression (Be a Mom Coping with Depression) by integrating face-to-face sessions with the web-based program Be a Mom.

The RCT will be a two-arm trial. Women who have had a child during the prior 12 months will be enrolled in the study. A minimum number of 110 women will be enrolled in the study. After agreeing to participate in the study, women will be screened and evaluated for the presence of clinically significant depressive symptoms (according to DSM-5) by a researcher (licensed psychologist). Participants who meet the eligibility criteria will be randomly assigned to one of the conditions: the blended intervention (Be a Mom Coping with Depression) or the control condition (online intervention - Be a Mom). The sample will be recruited online.

Participation in this study will last 6 months. The blended intervention will last about 3 months. Participants in both conditions will be invited by the researchers via email to complete baseline, post-intervention and follow-up (3-months post-intervention) assessments. Assessments will include self-report questionnaires to assess several indicators (e.g., depressive and anxiety symptoms, quality of life, marital satisfaction, mother-child bonding, and maternal self-efficacy), mechanisms that may be involved in the treatment response (e.g., psychological flexibility, emotional regulation, and self-compassion) and user's acceptability and satisfaction.

DETAILED DESCRIPTION:
In the present study, a blended intervention to treat postpartum depression (Be a Mom Coping with Depression) will be tested.

The main goal of this research is to apply and evaluate the acceptability and effectiveness of a blended cognitive-behavioral intervention for the treatment of postpartum depression by integrating face-to-face sessions with the web-based program Be a Mom. The efficacy of the intervention will be assessed considering two indicators: a) decrease or absence of clinically significant depressive symptoms at post-intervention and follow-up; and b) post-intervention and follow-up improvements in mother's psychosocial adjustment indicators (e.g., anxiety symptoms, marital satisfaction, maternal self-efficacy). The present study will also aim to investigate the mechanisms explaining the treatment response (e.g., psychological flexibility, self-compassion) and characteristics moderating the treatment response (e.g., motivation for therapy, therapeutic relationship).

The research design of the trial followed the methodological recommendations for the development and evaluation of blended interventions. A feasibility study was conducted prior to the randomized controlled trial (RCT), in order to evaluate preliminary version of the blended intervention. The feasibility study was conducted with women with a clinical diagnosis of postpartum depression according to the Structured Clinical Interview for DSM-5 (SCID-5) disorders criteria. Pre- and post-intervention assessments, using self-report questionnaires, and individual interviews were used to gather information concerning acceptability (relevance of contents and structure), feasibility, usability and preliminary clinical effectiveness (non-controlled). Appropriate adjustments to the blended protocol were carried out considering the results.

The RCT will be a two-arm trial. The intervention condition (blended intervention - Be a Mom Coping with Depression) will be compared with a control condition (online intervention - Be a Mom). The sample will include adult women who delivered an healthy baby in the postpartum period (up to 12 months postpartum). Women will be enrolled through online recruitment. A minimum number of 45 women per condition will be required (N=90). Accounting for the 20% of expected attrition rate over time, an anticipated sample of 110 women will be enrolled in the study.

Women who demonstrate interest in the study will be informed of the study goals, the structure and arms of the research and the researchers' and participants' roles. Women who agree to participate in the study will sign an informed consent form. All ethical requirements for research with humans are guaranteed.

After women's agreement to participate in the study, women who have a positive screen (indicating the presence of clinically relevant depressive symptoms) and meet the remaining eligibility criteria, will be interviewed (SCID-5) by the researcher (licensed psychologist) to assess the presence of clinically significant depressive symptoms. Women who do not fulfill the eligibility criteria will end their participation in the study and will be referred to intervention by local providers. Participants presenting at least 4 symptoms of a major depressive episode according to DSM-5, being one depressed mood or lost of pleasure or interest, with will be randomly assigned (blocked randomization, with allocation concealment) to one of the conditions: the intervention (blended intervention) or the control condition (online intervention).

Participation in this study will last 6 months. The blended Be a Mom intervention will last about 3 months and will be conducted by the researcher (licensed psychologist). Participants in both conditions will be invited by the researchers via email to complete baseline, post-intervention and follow-up (3-months post-intervention) assessments. Assessments will include self-report questionnaires to assess several indicators (e.g., depressive and anxiety symptoms, quality of life, marital satisfaction, mother-child bonding, and maternal self-efficacy), mechanisms that may be involved in the treatment response (e.g., psychological flexibility, emotional regulation, and self-compassion), and user's acceptability and satisfaction. The necessary statistical analyses will be conducted, using the intention-to-treat and per-protocol principles.

ELIGIBILITY:
Inclusion Criteria:

* Having 18 years or more;
* Being female;
* Being Portuguese;
* Baby's age up to 12 months;
* Presence of at least 4 symptoms of a major depressive episode according to DSM-5, being one depressed mood or lost of pleasure or interest;
* Having had a live healthy birth, with both woman and the child discharged from hospital;
* Internet and computer access;
* Being able to write and read Portuguese.

Exclusion Criteria:

* Presence of psychiatric comorbidity requiring alternative treatment primary to depression treatment (e.g., substance abuse, bipolar disorder);
* Presence of serious suicidal ideation;
* Presence of serious medical condition (either the participant or the baby);
* Currently receiving psychological or psychiatric treatment for depressive symptoms (antidepressant medication is allowed if stabilized for the last 3 months);
* Language difficulties that impede comprehension/reading-writing.

All participants will be informed that they will be randomized to one of the study groups and that will only be included if they give informed consent to participate in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in depressive symptoms | Baseline, 3 and 6 months
  Measured with Edinburgh Postnatal Depression Scale (EPDS). The total score can range between 0 and 30, and higher scores are indicative of more severe depressive symptoms.

SECONDARY OUTCOMES:
Changes from baseline in anxiety symptoms | Baseline, 3 and 6 months
  Measured with Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS). The total score for this subscale can range between 0 and 21, and higher scores indicate more anxiety symptomatology.
Changes from baseline in quality of life | Baseline, 3 and 6 months
  Measured with the Euroqol Five Dimension Scale (EQ-5D). The total score is obtained through an algorithm (the digits of the answers to the five dimensions) and it describes the health state.
Changes from baseline in the frequency of negative thoughts | Baseline, 3 and 6 months
  Measured with the Postnatal Negative Thoughts Questionnaire (PNTQ). The total score can range between 0 and 51, and higher scores indicate higher frequency of postpartum negative thoughts.
Changes from baseline in marital satisfaction | Baseline, 3 and 6 months
  Measured with the Satisfaction Subscale of the Investment Model Scale (IMS). The total score can range between 0 and 60, and higher scores indicate higher satisfaction with the relationship.
Changes from baseline in maternal self-efficacy | Baseline, 3 and 6 months
  Measured with the Perceived Maternal Parenting Self-Efficacy Questionnaire (PMP S-E). The total score can range between 20 and 80, and higher scores are indicative of higher perceived maternal self-efficacy.
Changes from baseline in mother-child bonding | Baseline, 3 and 6 months
  Measured with the Postpartum Bonding Questionnaire (PBQ). The total score can range between 0 and 60, and higher scores are indicative of a more impaired mother-child bond.
Changes from baseline in self-compassion | Baseline, 3 and 6 months
  Measured with the Self-Compassion Scale - Short Form (SCS-SF). The total score ranges between 1 and 48, and higher scores indicate higher levels of self-compassion.
Changes from baseline in emotional regulation | Baseline, 3 and 6 months
  Measured with the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF). The total score can range between 18 and 90, and higher scores are indicative of more difficulties in emotion regulation.
Changes from baseline in psychological flexibility | Baseline, 3 and 6 months
  Measured with the Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT). The total score can range between 0 and 108, and higher scores are indicative of higher scores are indicative of higher psychological flexibility.
Changes from baseline in expectancy for therapy | Baseline and 3 months
  Measured with the Credibility/Expectancy Questionnaire (CEQ). Higher scores indicate greater treatment credibility and expectations.
Therapeutic relationship | 3 months
  Measured with the Working Alliance Inventory - Short Revised (WAI-SR). The total score can range between 12 and 60, and higher scores indicate better therapeutic alliance.
Acceptability of the intervention for postpartum women | 3 months
  Measured through specific questions (to be developed by the researchers) to assess acceptability.
Usability of the intervention for postpartum women | 3 months
  Measured through specific questions (to be developed by the researchers) to assess usability.
Feasibility of the online program for postpartum women as measured by number of website logins | 3 months
  Measured through the number of user's website logins.
Feasibility of the program for postpartum women as measured by website average visit length | 3 months
  Measured through the number of user's website average visit length.
Feasibility of the intervention for postpartum women as measured by dropout rate | 3 months
  Measured through the number of participants that dropped out from the intervention before completing it.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology and Education Sciences, University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
After the conclusion of the trial, the investigators plan to share the results of the study both with scientific community and health professionals.

REFERENCES:
- [Derived] Branquinho M, Canavarro MC, Fonseca A. Blended CBT Intervention vs. a Guided Web-Based Intervention for Postpartum Depression: Results From a Pilot Randomized Controlled Trial. Clin Psychol Psychother. 2024 Nov-Dec;31(6):e70007. doi: 10.1002/cpp.70007. PMID 39500299